CLINICAL TRIAL: NCT00373438
Title: Randomized Clinical Trial in Order to Assess the Effect of Fetoscopic Tracheal Balloon Occlusion on the Postnatal Disease Course in Neonates With Left Congenital Diaphragmatic Hernia - FDH-ECMO/BALLOON-TRIAL
Brief Title: Fetoscopic Tracheal Balloon Occlusion in Left Diaphragmatic Hernia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Collaborators: Universitätsmedizin Mannheim (Other)
Responsible Party: Thomas Kohl MD, German Center for Fetal Surgery & Minimally-Invasive Therapy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDH-ECMO/BALLOON-TRIAL-135/06; 135/06
Record Dates: First submitted 2006-09-06; First posted 2006-09-08 (Estimated); Last update posted 2009-01-06 (Estimated); Status verified 2009-01

CONDITIONS: Diaphragmatic Hernia
Keywords: Congenital diaphragmatic hernia; tracheal occlusion; fetus; fetal surgery; fetoscopy; ECMO
MeSH Terms: conditions — Hernia, Diaphragmatic; Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (No Intervention)
  Interventions: Procedure: Fetoscopic tracheal balloon occlusion
- B (Experimental): Fetoscopic tracheal occlusion
  Interventions: Procedure: Fetoscopic tracheal balloon occlusion

INTERVENTIONS:
Procedure: Fetoscopic tracheal balloon occlusion — Maternal local anesthesia, percutaneous ultrasound-guided fetal analgo-sedation and relaxation, percutaneous ultrasound-guided access into amniotic cavity with trocar, fetoscopic tracheal ballon occlusion, removal of fetoscope and trocar, maternal abdominal closure, skin-to-skin time 30 minutes

SUMMARY:
Left diaphragmatic hernia detected during fetal life carries a high risk for postnatal lung failure due to lung underdevelopment and pulmonary hypertension. In severe cases, extracorporeal membrane oxygenation (ECMO) is used as a life-saving intensive care means to enable survival of severely affected infants.

Clinical experience from prospective controlled non-randomized case series with fetoscopic tracheal balloon occlusion has seen improved survival rates in contrast to untreated controls.

Therefore, the purpose of this randomized clinical trial in a less severely affected subgroup of patients is whether by fetoscopic tracheal occlusion, the intensity of postnatal intensive care therapy might be reduced. Primary outcome measure is the need for postnatal ECMO therapy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women from European countries carrying fetuses with left diaphragmatic hernia.
* Normal karyotype, no further severe anomalies on prenatal ultrasound study.
* Fetal liver herniation into the chest; gestational age-related lung volume between 20-25% of normal as determined by magnetic resonance imaging between 30+0 - 34+0 weeks+days of gestation.

Exclusion Criteria:

* Any maternal disease or condition that would result in an increased risk to her health from the experimental procedure.
* Abnormal fetal karyotype, further severe fetal anomalies on prenatal ultrasound.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2009-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Need for postnatal ECMO therapy | First two days of life

SECONDARY OUTCOMES:
Survival to discharge from hospital | Days to discharge
Maternal morbidity | Until maternal discharge
Fetal / Neonatal morbidity | Overall & at discharge from hospital
Premature preterm rupture of membranes | Following the interventions over the remainder of gestation
Unintended preterm delivery | Following the interventions before scheduled elective delivery
Days in intensive care | Number of day until discharge from ICU
Days in hospital | Number of days until discharge from hospital
Oxygen dependency on discharge | Days until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kohl, MD, Principal Investigator — German Center for Fetal Surgery & Minimally-Invasive Therapy, University of Bonn, Germany; Thomas Schaible, MD, Principal Investigator — Neonatal Intensive Care Unit (ECMO center), University of Mannheim, Germany
Locations (1):
- German Center for Fetal Surgery & Minimally Invasive Therapy, Bonn, Germany

REFERENCES:
- [Background] Kohl T, Gembruch U, Filsinger B, Hering R, Bruhn J, Tchatcheva K, Aryee S, Franz A, Heep A, Muller A, Bartmann P, Loff S, Hosie S, Neff W, Schaible T; German Center for Fetal Surgery Diaphragmatic Hernia Task Group. Encouraging early clinical experience with deliberately delayed temporary fetoscopic tracheal occlusion for the prenatal treatment of life-threatening right and left congenital diaphragmatic hernias. Fetal Diagn Ther. 2006;21(3):314-8. doi: 10.1159/000091363. PMID 16601345